CLINICAL TRIAL: NCT06017609
Title: A Phase 2a, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy, Safety and Tolerability of JTT-861 Administered for 12 Weeks in Subjects With Heart Failure With Reduced Ejection Fraction
Brief Title: Evaluate Efficacy, Safety and Tolerability of JTT-861 in Subjects With Heart Failure With Reduced Ejection Fraction
Acronym: POWER-HF
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Akros Pharma Inc. (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AT861-G-22-002
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Chronic Heart Failure
Keywords: JTT-861; Efficacy; Safety; Tolerability; Chronic Heart Failure; HFrEF; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- JTT-861 Dose 1 (Experimental): JTT-861 Capsules Dose 1 orally once daily for 12 weeks
  Interventions: Drug: JTT-861 Capsules
- JTT-861 Dose 2 (Experimental): JTT-861 Capsules Dose 2 orally once daily for 12 weeks
  Interventions: Drug: JTT-861 Capsules
- Placebo (Experimental): Placebo Capsules orally once daily for 12 weeks
  Interventions: Drug: Placebo Capsules

INTERVENTIONS:
Drug: JTT-861 Capsules — Active drug capsules containing JTT-861
  Arms: JTT-861 Dose 1; JTT-861 Dose 2
Drug: Placebo Capsules — Placebo capsules matching in appearance to the active drug capsules
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy, safety, tolerability and pharmacokinetics of JTT-861 administered once daily for 12 weeks in subjects with heart failure with reduced ejection fraction (HFrEF) who are on a stable, guideline-directed medical therapy for heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Has a clinical diagnosis of symptomatic heart failure (HF) ≥90 days prior to the Screening Visit;
* Is in New York Heart Association (NYHA) functional class II or III at the Screening Visit;
* Is on stable, guideline-directed therapy for HF, consistent with American Heart Association (AHA), American College of Cardiology (ACC), Heart Failure Society of America (HFSA) or European Society of Cardiology (ESC) guidelines for ≥4 weeks prior to the Screening Visit (with at least half of maximal labeled dose of renin-angiotensin-aldosterone system (RAAS) inhibitors and β-blockers, if tolerated);
* Has left ventricular ejection fraction (LVEF) ≤35% at the Screening Visit;
* Has a serum N-terminal pro b-type natriuretic peptide (NT-pro-BNP) level ≥600 pg/mL (or ≥900 pg/mL if the subject has atrial fibrillation or atrial flutter) at the Screening Visit.

Exclusion Criteria:

* Has a confirmed acute myocardial infarction (MI) (i.e., Type 1) or unstable angina within 90 days prior to the Screening Visit;
* Has a history of coronary revascularization (percutaneous coronary intervention [PCI] and/or coronary artery bypass graft [CABG]) or other cardiovascular surgery within 90 days prior to the Screening Visit or planned cardiovascular surgery during the study through the Follow-up Visit);
* Has started cardiac resynchronization therapy (CRT) within 90 days prior to the Screening Visit or has planned CRT during the study through the Follow-up Visit;
* Has clinically significant congenital heart disease, active myocarditis or constrictive pericarditis;
* Has current acute decompensated HF requiring additional treatment with diuretics, vasodilators and/or inotropic medications at the Screening Visit;
* Has clinically significant chronic renal insufficiency (i.e., estimated glomerular filtration rate [eGFR] <30 mL/min/1.73 m2 calculated by the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] creatinine equation) at the Screening Visit.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to end of treatment (EOT) in left ventricular ejection fraction (LVEF) as assessed by two-dimensional echocardiography (2D-echo) | 12 Weeks
Change from baseline to EOT in left ventricular end-systolic volume (LVESV) index as assessed by 2D-echo | 12 Weeks
Change from baseline to EOT in left ventricular end-diastolic volume (LVEDV) index as assessed by 2D-echo | 12 Weeks
Change from baseline to EOT in left atrial volume (LAV) as assessed by 2D-echo | 12 Weeks
Change from baseline to EOT in N-terminal pro b-type natriuretic peptide (NT-pro-BNP) values | 12 Weeks
Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) scores from baseline | 16 Weeks
  General Scoring Guideline: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent
Number of subjects with treatment-emergent adverse events | Up to 16 Weeks
Trough plasma concentrations of JTT-861 | Weeks 4, 8 and 12
Post-dose plasma concentrations of JTT-861 | Weeks 2, 4 and 8

CONTACTS AND LOCATIONS:
Locations (74):
- United States (20):
  - Arensia Exploratory Medicine Inc., Phoenix, Arizona
  - Nature Coast Clinical Research, Crystal River, Florida
  - Indago Research & Health Center, Inc., Hialeah, Florida
  - Med Research of Florida, Miami, Florida
  - Pharma Medical Innovation, Inc., Miami Lakes, Florida
  - Floridian Clinical Research, Miami Lakes, Florida
  - Affinity Health, Park Ridge, Illinois
  - ASHA Clinical Research-Munster, LLC, Hammond, Indiana
  - Monroe Research, LLC, West Monroe, Louisiana
  - Henry Ford Hospital, Detroit, Michigan
  - Profound Research LLC, Farmington Hills, Michigan
  - NextStage Clinical Research - (Kansas City [01]), Kansas City, Missouri
  - Laurelton Heart Specialist P.C., Rosedale, New York
  - Capital Area Research, LLC, Camp Hill, Pennsylvania
  - Onsite Clinical Solutions, LLC, Rock Hill, South Carolina
  - NextStage Clinical Research-Beaumont- (01), Beaumont, Texas
  - Cypress Heart and Vascular Center, Cypress, Texas
  - NextStage Clinical Research-Port Arthur-(02), Port Arthur, Texas
  - Sherman Clinical Research, Sherman, Texas
  - Waco Cardiology Associates - NextStage Clinical Research, Waco, Texas
- Bulgaria (11):
  - Ambulatory for Specialized Outpatient Medical Care in Cardiology Individual Practice- Dr. Elena Dotcheva EOOD, Burgas
  - Multiprofile Hospital for Active Treatment "Ivan Skenderov", Gotse Delchev
  - Multiprofile Hospital For Active Treatment Ivan Skenderov EOOD, Gotse Delchev
  - University Multiprofile Hospital for Active Treatment Georgi Stranski, EAD, Pleven
  - Multiprofile Hospital For Active Treatment Heart and Brain EAD, Pleven
  - University Multiprofile Hospital For Active Treatment Saint Georgi EAD, Plovdiv
  - Acibadem City Clinic University Multiprofile Hospital For Active Treatment EOOD, Sofia
  - Medical Center Hera EOOD, Sofia
  - Multiprofile Hospital for Active Treatment Tsaritsa Yoanna - ISUL EAD, Sofia
  - Diagnostic Consultative Center Convex EOOD, Sofia
  - University Multiprofile Hospital for Active Treatment. Sv Anna - Sofia AD, Sofia
- Czechia (9):
  - MUDr. Libor Nechvatal s.r.o., Brno
  - Centrum pro zdraví, s.r.o., Brno
  - Vojenská nemocnice Brno, Brno
  - Fakultní nemocnice Brno, Brno
  - Edumed s.r.o., Broumov
  - Edumed s.r.o., Hradec Králové
  - Edumed s.r.o., Jaroměř
  - Edumed s.r.o., Náchod
  - Fakultní nemocnice Ostrava, Ostrava-Poruba
- Poland (11):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - American Heart of Poland S.A., Chrzanów
  - American Heart of Poland S.A., Dąbrowa Górnicza
  - Kardio Brynów Sp. z o.o., Katowice
  - Centrum Rehabilitacji I Kardiologii Solutaris Prokopczuk Sp.j., Kędzierzyn-Koźle
  - Wojewodzki Specjalistyczny Szpital Im Dr Wl Bieganskiego, Lodz
  - Uniwersytecki Szpital Kliniczny Nr 4 w Lublinie, Lublin
  - Trialmed CRS Piotrków Trybunalski, Piotrkow Trybunalski
  - NZOZ "Pro Cordis" Sopockie Centrum Badań Kardiologicznych Paweł Miękus, Sopot
  - American Heart of Poland S.A., Tychy
  - 4 Wojskowy Szpital Kliniczny z Polikliniką Samodzielny Publiczny Zakład Opieki Zdrowotnej we Wrocławiu, Wroclaw
- Romania (11):
  - Thera Card S.R.L, Brasov
  - Spitalul Clinic Judetean De Urgenta Brasov, Brasov
  - Spitalul Clinic De Urgență Sf. Pantelimon București, Bucharest
  - Spitalul Universitar de Urgență București, Bucharest
  - Mat Cord Biomedica SRL, Buzău
  - Angiocare S.R.L., Cluj-Napoca
  - Cardio Med SRL, Craiova
  - Spitalul Clinic Județean de Urgență Craiova, Craiova
  - Cardio Med SRL, Târgu Mureş
  - CMI Dr. Podoleanu Cristian, Târgu Mureş
  - Spitalul Clinic Municipal de Urgenţă Timişoara, Timișoara
- Spain (12):
  - Hospital Clínico Universitario de Santiago, A Coruña
  - Hospital del Mar - Parc de Salut Mar, Barcelona
  - Area Sanitaria De Ferrol - Hospital Arquitecto Marcide, Ferrol
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No